CLINICAL TRIAL: NCT03233854
Title: Phase 1 Dose Escalation Study of CD19/CD22 Chimeric Antigen Receptor (CAR) T Cells With or Without NKTR-255 in Adults With Recurrent or Refractory B Cell Malignancies
Brief Title: CD19/CD22 Chimeric Antigen Receptor (CAR) T Cells With or Without NKTR-255 in Adults With Recurrent or Refractory B Cell Malignancies
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-41382; NCI-2017-01291 (Registry Identifier: National Cancer Institute Clinical Trials Reporting Program)
Record Dates: First submitted 2017-07-26; First posted 2017-07-31 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: B Acute Lymphoblastic Leukemia; CD19 Positive; Minimal Residual Disease; Philadelphia Chromosome Positive
MeSH Terms: conditions — Burkitt Lymphoma; Neoplasm, Residual | interventions — Immunotherapy, Adoptive; Cyclophosphamide; fludarabine phosphate; NKTR-255

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (CD19/CD22 CAR T cells, chemotherapy, NKTR-255) (Experimental): Patients receive cyclophosphamide IV over 60 minutes and fludarabine phosphate IV over 30 minutes on days -5 to -3. Patients then receive CD19/CD22 CAR T cells IV over 10-20 minutes on day 0. On Day 14 after CAR-T, eligible patients will be given NKTR-255 IV over 30 minutes, and it will be repeated every 28 days for up to 6 cycles. Patients that benefited from the first dose of CD19/CD22 CAR T cells, had no unacceptable side effects, and have enough cells left over may receive 2 or 3 additional doses of CD19/CD22 CAR T cells.
  Interventions: Biological: Chimeric Antigen Receptor T-Cell Therapy; Drug: Cyclophosphamide; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration; Drug: NKTR-255

INTERVENTIONS:
Biological: Chimeric Antigen Receptor T-Cell Therapy — Given CD19/CD22 CAR T cells IV
  Other Names: CAR T-cell therapy
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Questionnaire Administration — Ancillary studies
Drug: NKTR-255 — Given IV

SUMMARY:
This phase I trial studies the side effects of CD19/CD22 chimeric antigen receptor (CAR) T cells when given together with chemotherapy and NKTR-255, and to see how well they work in treating patients with CD19 positive B acute lymphoblastic leukemia that has come back or does not respond to treatment. A CAR is a genetically-engineered receptor made so that immune cells (T cells) can attack cancer cells by recognizing and responding to the CD19/CD22 proteins. These proteins are commonly found on diffuse large B-cell lymphoma and B acute lymphoblastic leukemia. Drugs used in chemotherapy, such as cyclophosphamide and fludarabine phosphate, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. NKTR-255 is an investigational IL-15 receptor agonist designed to boost the immune system's natural ability to fight cancer. Giving CD19/CD22-CAR T cells and chemotherapy in combination with NKTR-255 may work better in treating patients with diffuse large B-cell lymphoma or B acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the feasibility of producing CD19/CD22 CAR T cells meeting the established release criteria.

II. Assess the safety of administering escalating doses of autologous CD19/CD22 CAR T cells that meet established release specifications in adults with B cell hematologic malignancies following a cyclophosphamide/fludarabine conditioning regimen.

III. Assess the safety and feasibility of administering repeated doses of NKTR-255 intravenously after CD19/CD22-CAR T cell infusions in adults with ALL using a dose escalation design.

IV. Determine the recommended phase 2 dose (RP2D) of NKTR-255 when administered following CD19/CD22-CAR T cell infusion in adults with ALL

SECONDARY OBJECTIVES:

I. Evaluate the ability of CD19/CD22 CAR T cells to mediate clinical activity in adults with DLBCL and adults with ALL.

II. Characterize the pharmacokinetics (PK) of NKTR-255 when administered post CD19/CD22 CAR T cell infusion.

III. Explore the rate of relapse, progression free survival (PFS) and overall survival (OS) in subjects receiving CD19/CD22 CAR T cells, followed by up to 6 cycles of NKTR-255

ELIGIBILITY:
For B acute lymphoblastic leukemia (ALL)

1. Confirmed diagnosis of relapsed or refractory B-cell ALL of one of the following types:

   * Chemotherapy refractory disease in subjects with B-ALL, defined as progression or stable disease after one line of therapy.
   * Recurrence of disease after achieving CR.
2. Subjects with persistent or relapsed minimal residual disease (MRD) (by flow cytometry, PCR, FISH, or next generation sequencing) require verification of MRD positivity on two occasions at least 4 weeks apart.
3. Subjects with Philadelphia Chromosome positive acute lymphoblastic leukemia (Ph+ALL) subjects are eligible if they progressed after receiving a tyrosine kinase inhibitor (TKI).
4. Subjects with recurrence of isolated CNS relapse after achieving complete remission (CR); if relapsed with MRD, will require verification of MRD positivity on two occasions at least 4 weeks apart.
5. CD19 positive expression- CD19 expression is required at any time since diagnosis. If patient has received anti-CD19 targeted therapy (i.e. Blinatumomab or CD19-CAR T cells), then CD19 expression must be subsequently demonstrated. CD19 expression may be detected by immunohistochemistry or by flow cytometry. The choice of whether to use flow cytometry or immunohistochemistry will be determined by what is the most easily available tissue sample in each subject. In general, immunohistochemistry will be used for lymph node biopsies, flow cytometry will be used for peripheral blood and bone marrow samples.
6. Subjects who have undergone autologous SCT with disease progression or relapse following SCT are eligible. Subjects who have undergone allogeneic SCT will be eligible if, in addition to meeting other eligibility criteria, they have elelino evidence of GVHD and have been without immunosuppressive agents for at least 30 days.
7. Subjects who have undergone prior anti-CD19 or anti-CD22 CAR therapy must be at least 30 days post CAR infusion and may not have eficence of persistnce of CAR T cells in blood smples (circulating levels of genetically modified cels of >/= 5% by flow cytometry.
8. Must have evaluable or measurable disease. Lesions that have been previously irradiated will be considered measurable only if progression has been documented following completion of radiation therapy.
9. At least 2 weeks or 5 half-lives, whichever is shorter, must have elapsed since any prior systemic therapy at the time the subject is planned for leukapheresis, except for systemic inhibitory/stimulatory immune checkpoint therapy, which requires 5 half-lives.

   Exceptions:
   1. There is no time restriction with regard to prior intrathecal chemotherapy (incl. steroids) provided there is complete recovery from any acute toxic effects;
   2. Subjects who are on standard ALL maintenance type chemotherapy (vincristine, 6-mercaptopurine or oral methotrexate) may be enrolled provided that chemotherapy is discontinued at least 1 week or 5 half-lives (whichever is shorter) prior to apheresis.
   3. Subjects receiving steroid therapy at physiologic replacement doses (≤5 mg/day of prednisone or equivalent doses of other corticosteroids) only are allowed provided there has been no increase in dose for at least 2 weeks prior to starting apheresis;
   4. For radiation therapy: Radiation therapy must have been completed at least 3 weeks prior to apheresis, with the exception that there is no time restriction if the volume of bone marrow treated is less than 10% and also the subject has measurable/evaluable disease outside the radiation port.
10. Toxicities due to prior therapy must be stable and recovered to ≤ Grade 1 (except for clinically non-significant toxicities such as alopecia)
11. Age 18 or older
12. Eastern cooperative oncology group (ECOG) performance status of 0, 1, or 2; or Karnofsky ≥ 60%
13. Normal Organ and Marrow Function (supportive care is allowed per institutional standards, i.e. filgrastim, transfusion)

    1. ANC ≥ 1000/uL*
    2. Platelet count ≥ 50,000/uL*
    3. Absolute lymphocyte count ≥ 300/uL*
    4. Adequate renal, hepatic, pulmonary and cardiac function defined as:
    5. Creatinine ≤ 2 mg/dL or creatinine clearance ≥ 60 mL/min
    6. Serum ALT or AST ≤ 5x ULN (Elevated ALT/AST associated with leukemia or lymphoma involvement of the liver will not disqualify a subject; only one value required for eligibility).
    7. Total bilirubin ≤ 1.5 mg/dl, except in subjects with Gilbert's syndrome.
    8. Cardiac ejection fraction ≥ 45%, no evidence of physiologically significant pericardial effusion as determined by an ECHO, MUGA or Cardiac MRI [performed within 180 days or after most recent anthracycline based treatment or mediastinal radiation therapy (whichever is most recent)]
    9. No clinically significant ECG findings
    10. No clinically significant pleural effusion
    11. Baseline oxygen saturation > 92% on room air * A subject will not be excluded because of cytopenia if it is felt by the investigator to be due to underlying leukemia/lymphoma.
14. Subjects with CNS involvement are eligible as long as there are no overt signs or symptoms that in the evaluation of the investigator would mask or interfere with the neurological assessment of toxicity.
15. Females of childbearing potential must have a negative serum or urine pregnancy test (females who have undergone surgical sterilization or who have been postmenopausal for at least 2 years are not considered to be of childbearing potential)
16. Subjects of child-bearing or child-fathering potential must be willing to practice birth control from the time of enrollment on this study and for four (4) months after receiving the preparative lymphodepletion regimen or 1 month after the last dose of NKTR_255, whichever is later.
17. Ability to give informed consent. Must be able to give informed consent. Subjects unable to give informed consent will not be eligible for this study.

=ELIGIBILITY TO RECEIVE NKTR-255=

* Received a CD19/CD22 CAR-T infusion
* No persisting grade ≥1 CRS or greater than grade 1 fever within 12 hours preceding NKTR-255 infusion
* No grade 4 CRS within 96 hours preceding NKTR-255 infusion
* No persisting grade ≥ 2 neurotoxicity on the day of NKTR-255 infusion
* No previous grade ≥ 3 neurotoxicity of > 48 hours duration at any time preceding NKTR-255 infusion
* ANC ≥ 1000/µL
* No intervention with tocilizumab and/or dexamethasone within 48 hours preceding NKTR-255 infusion
* No active, serious, and uncontrolled infection(s)
* No contraindications according to the PI's assessment
* Life expectancy > 30 days

Exclusion Criteria:

1. History of other malignancy, unless disease free for at least 3 years. At the discretion of the Principal Investigator, subjects in remission for 1-2 years prior to enrollment may be deemed eligible after considering the nature of other malignancy, likelihood of recurrence during one year following CAR therapy, and impact of prior treatment on risk of CD19/CD22-CAR T cells. Subjects in remission <1 year are not eligible.

   * Exception: Nonmelanoma skin cancer or carcinoma in situ (e.g. cervix, bladder, breast) is eligible.
   * Hormonal therapy in subjects in remission >1 year will be allowed.
2. Presence of fungal, bacterial, viral, or other infection that is uncontrolled. Simple UTI and uncomplicated bacterial pharyngitis are permitted if responding to active treatment.
3. Known history of infection with any of the following:

   * HIV
   * Hepatitis B (HBsAg positive)
   * Hepatitis C virus (anti-HCV positive) A history of hepatitis B or hepatitis C is permitted if the viral load is undetectable per quantitative PCR and/or nucleic acid testing.
4. Presence of a seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement that in the judgment of the investigator may impair the ability to evaluate neurotoxicity.
5. History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, or other clinically significant cardiac disease within 12 months of enrollment
6. Any medical condition that in the judgement of the investigator is likely to interfere with assessment of safety or efficacy of study treatment
7. History of severe immediate hypersensitivity reaction to any of the agents used in this study
8. Women who are pregnant or breastfeeding
9. In the investigator's judgment, the subject is unlikely to complete all protocol-required study visits or procedures, including follow-up visits, or comply with the study requirements for participation.
10. Previous treatment with interleukin-2 or interleukin-15.
11. Confirmed diagnosis of relapsed/refractory biphenotypic BT cell ALL
12. Primary immunodeficiency or history of autoimmune disease (e.g. Crohns, rheumatoid arthritis, systemic lupus) requiring systemic immunosuppression/systemic disease modifying agents within the last 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2035-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of dose limiting toxicities (DLTs) following chemotherapy preparative regimen and infusion of CD19/CD22 chimeric antigen receptor (CAR) T cells | Up to 28 days
  Safety data will be analyzed per standard methods and interpreted descriptively for each dose cohort. Safety data will be summarized for each dose cohort separately and for all dose cohorts combined. Adverse events will be assessed using the CTCAE version 4.03 for type and severity of event. Serious Adverse Events will be summarized for each dose cohort and for all dose cohorts combined. Reasons for discontinuation of study therapy will be tabulated.
Maximum tolerated dose of CD19/CD22 chimeric antigen receptor (CAR) T cells defined as the dose level immediately below the level at which the enrollment is stopped due to a dose limiting toxicity | Up to 28 days
  Will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Rate of successful manufacture and expansion of the CD19/CD22 chimeric antigen receptor (CAR) T cells to satisfy the targeted dose level and meet the required release specifications outlined in the Certificate of Analysis | Up to 15 years
  In addition to aiming to evaluate up to 6 subjects at a given dose level with respect to toxicity, the number of subjects which can successfully manufacture the targeted dose number will be determined.

SECONDARY OUTCOMES:
Overall survival | From the start of the preparative regimen until death, assessed for up to 15 years
  Will be assessed by dose cohort.
Progression free survival | From the start of the preparative regimen until the documentation of disease progression or death due to any cause, whichever occurs first, assessed for up to 15 years
  Will be assessed by dose cohort.
The ability to achieve a clinical response after administration of CD19/CD22 chimeric antigen receptor (CAR) T cells | Up to 15 years
  Will be assessed by the Response Criteria for Lymphoma and the Response Criteria for Acute Lymphoblastic Leukemia.

OTHER OUTCOMES:
Alterations in early B cell development induced by immune pressure exerted via CD19/CD22 chimeric antigen receptor (CAR) T cells | Up to 15 years
  Will be evaluated.
CD19/CD22 chimeric antigen receptor (CAR) T cell properties | Up to 15 years
  Will explore correlations with CAR T cell efficacy and persistence.
Establish the utility of chromatin structure and epigenomic technology to characterize chimeric antigen receptor (CAR) T cell therapies | Up to 15 years
  Investigators will attempt to establish parameters for how best to utilize the technology in CAR research to: establish basis for blood therapeutic monitoring; derive blood biomarkers for prediction of the safety and efficacy of CAR cell therapy; and develop metrics for CAR T product release criteria that can be used during the manufacturing of the product.
Frequency of CD22+ expression on leukemia cells | Up to 15 years
  Will correlate with clinical response to CAR T cells.
Persistence of CD19/CD22 chimeric antigen receptor (CAR) T cells blood, bone marrow, and cerebral spinal fluid | Up to 15 years
  Will be assessed by flow cytometry. Will be analyzed and reported as time from T cell infusion.
Relapse with loss or diminished expression of CD19, CD22 and/or NKTR-255 | Up to 15 years
  Will be evaluated.
Immunogenicity of NKTR-255 | Up to 15 years
  Will be evaluated when administered post CD19/CD22 CAR T cell infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Lori Muffly, MD, MS, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Srinagesh H, Jackson C, Shiraz P, Jeyakumar N, Hamilton M, Egeler E, Mavroukakis S, Kuo A, Cancilla J, Sahaf B, Agarwal N, Kanegai A, Kramer AM, Arai S, Bharadwaj S, Dahiya S, Hosoya H, Johnston L, Kennedy V, Liedtke M, Lowsky R, Mikkilineni L, Negrin R, Rezvani A, Sidana S, Shizuru J, Smith M, Weng WK, Feldman S, Frank MJ, Lee Z, Tagliaferri M, Marcondes AM, Miklos D, Mackall C, Muffly L. A phase 1 clinical trial of NKTR-255 with CD19-22 CAR T-cell therapy for refractory B-cell acute lymphoblastic leukemia. Blood. 2024 Oct 17;144(16):1689-1698. doi: 10.1182/blood.2024024952. PMID 38968138
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338
- [Derived] Spiegel JY, Patel S, Muffly L, Hossain NM, Oak J, Baird JH, Frank MJ, Shiraz P, Sahaf B, Craig J, Iglesias M, Younes S, Natkunam Y, Ozawa MG, Yang E, Tamaresis J, Chinnasamy H, Ehlinger Z, Reynolds W, Lynn R, Rotiroti MC, Gkitsas N, Arai S, Johnston L, Lowsky R, Majzner RG, Meyer E, Negrin RS, Rezvani AR, Sidana S, Shizuru J, Weng WK, Mullins C, Jacob A, Kirsch I, Bazzano M, Zhou J, Mackay S, Bornheimer SJ, Schultz L, Ramakrishna S, Davis KL, Kong KA, Shah NN, Qin H, Fry T, Feldman S, Mackall CL, Miklos DB. CAR T cells with dual targeting of CD19 and CD22 in adult patients with recurrent or refractory B cell malignancies: a phase 1 trial. Nat Med. 2021 Aug;27(8):1419-1431. doi: 10.1038/s41591-021-01436-0. Epub 2021 Jul 26. PMID 34312556